CLINICAL TRIAL: NCT02019914
Title: Effects of Continuous Positive Airway Pressure Therapy for Obstructive Sleep Apnea on PTSD Symptoms
Brief Title: Effects of CPAP Therapy on PTSD Symptoms
Status: Completed | Type: Observational
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H130095
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: PTSD; Sleep; Obstructive Sleep Apnea; Quality of Life
Keywords: PTSD; CPAP; OSA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PTSD and OSA: Veterans diagnosed with Post Traumatic Stress Disorder (PTSD) and Obstructive Sleep Apnea (OSA), interested in a trial of CPAP therapy.

SUMMARY:
The purpose of this study is to evaluate the effects of treating Obstructive Sleep Apnea (OSA) with continuous positive airway pressure (CPAP) therapy on symptoms of post traumatic stress disorder (PTSD). The study hypotheses are that CPAP use will improve PTSD symptoms overall and that CPAP use will improve sleep quality and duration, nocturnal symptoms related to PTSD, mood, daytime sleepiness, sleep-related quality of life, and general health perception.

DETAILED DESCRIPTION:
Post traumatic stress disorder (PTSD) is associated with increased healthcare utilization, decreased functional status, and overall poor health. Sleep disturbances in PTSD are common, including nightmares, dream enactment, and poor sleep quality. Obstructive sleep apnea (OSA) is also highly prevalent in the veteran population and may exacerbate PTSD symptoms by triggering arousals from sleep that promote recollection of dreams, enactment of dreams, and disrupt sleep continuity. Improvements in sleep quality and PTSD symptoms have been reported when OSA is treated with continuous positive airway pressure (CPAP) therapy. However, formal assessment using validated questionnaires and documentation of CPAP compliance to correlate with these tools has not yet been performed. This study will recruit veterans with PTSD who have been newly diagnosed with OSA and who are willing to try CPAP therapy. Baseline assessments of PTSD symptoms, daytime sleepiness, sleep-related quality of life, sleep quality, general health perception, and mood will be performed before initiation of treatment and after 3 and 6 months of therapy.

This study will have the following specific aims:

Aim 1: To evaluate the effect of CPAP use on PTSD symptoms.

Hypothesis: After 6 months of treatment, CPAP use will improve PTSD symptoms as assessed by the PTSD checklist (PCL-S).

Aim 2: To evaluate the effect of CPAP use on 1)sleep quality and duration, 2)nocturnal symptoms of nightmares, movement disorders, dream enactment, and insomnia, 3)mood, 4)daytime sleepiness, 5)sleep-related quality of life, and 6) general health perception.

Hypothesis: After 6 months of treatment, CPAP use will improve sleep quality, sleep duration, mood, daytime sleepiness, sleep-related quality of life, general health perception, and nocturnal symptoms of nightmares, movement disorders, dream enactment, and insomnia.

ELIGIBILITY:
Inclusion Criteria:The intent is to recruit a study population that is as representative as possible of the veteran PTSD population. Thus, entry criteria are as inclusive as possible:

* age >18 year
* confirmed diagnosis of PTSD (PCL checklist minimum score of 45)
* confirmed diagnosis of sleep apnea (apnea hypopnea index >5/h)
* newly starting CPAP (not previously treated)

Exclusion Criteria:

* fatal co-morbidity with life expectancy of less than 6 months,
* residing in a geographically remote area that would make follow up at 3 and 6 months difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with confirmed diagnoses of PTSD and OSA who are willing to try CPAP therapy.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms measured by the PTSD checklist (PCL-S). | Baseline, 3 months, 6 months
  A change of -10 points on the PCL-S has been previously determined to be clinically significant.

SECONDARY OUTCOMES:
Daytime Sleepiness measured by the Epworth Sleepiness Scale (ESS) | Baseline, 3 months, 6 months
Sleep Related Quality of life with be assessed using the Functional Outcomes of Sleep Questionnaire (FOSQ-10). | Baseline, 3 months, 6 months
  The FOSQ-10 consists of 10 questions, with a lower score indicating more difficulty with activity due to poor sleep.
Change in sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI). | Baseline, 3 months, 6 months
  This is a 19 item self-report assessment of sleep quality and degree of sleep difficulties over the past month. A global score>/=5 is considered poor sleep quality.
Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). | Baseline, 3 months, 6 months
  The PHQ-9 is a self report depression measure and is a quick, valid assessment of depression. Depression is a common comorbid condition with PTSD.
General health related quality of life. | Baseline, 3 months, 6 months
  This will be assessed using a likert scale question asking subjects to rate their quality of life for 2 preceding days based on spiritual, emotional, physical, social and financial aspects of their lives.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F Sarmiento, MD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Vasterling JJ, Schumm J, Proctor SP, Gentry E, King DW, King LA. Posttraumatic stress disorder and health functioning in a non-treatment-seeking sample of Iraq war veterans: a prospective analysis. J Rehabil Res Dev. 2008;45(3):347-58. doi: 10.1682/jrrd.2007.05.0077. PMID 18629744
- [Background] Kubzansky LD, Koenen KC, Spiro A 3rd, Vokonas PS, Sparrow D. Prospective study of posttraumatic stress disorder symptoms and coronary heart disease in the Normative Aging Study. Arch Gen Psychiatry. 2007 Jan;64(1):109-16. doi: 10.1001/archpsyc.64.1.109. PMID 17199060
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Hoge CW, Terhakopian A, Castro CA, Messer SC, Engel CC. Association of posttraumatic stress disorder with somatic symptoms, health care visits, and absenteeism among Iraq war veterans. Am J Psychiatry. 2007 Jan;164(1):150-3. doi: 10.1176/ajp.2007.164.1.150. PMID 17202557
- [Background] Kulka RA, Schlenger WA, Fairbanks JA, et al. Trauma and the Vietnam War generation: report of findings from the National Vietnam Veterans Readjustment Study (1990). New York: Brunner/Mazel.
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kang HK, Natelson BH, Mahan CM, Lee KY, Murphy FM. Post-traumatic stress disorder and chronic fatigue syndrome-like illness among Gulf War veterans: a population-based survey of 30,000 veterans. Am J Epidemiol. 2003 Jan 15;157(2):141-8. doi: 10.1093/aje/kwf187. PMID 12522021
- [Background] El-Sherbini AM, Bediwy AS, El-Mitwalli A. Association between obstructive sleep apnea (OSA) and depression and the effect of continuous positive airway pressure (CPAP) treatment. Neuropsychiatr Dis Treat. 2011;7:715-21. doi: 10.2147/NDT.S26341. Epub 2011 Dec 13. PMID 22247613
- [Background] Belleville G, Guay S, Marchand A. Impact of sleep disturbances on PTSD symptoms and perceived health. J Nerv Ment Dis. 2009 Feb;197(2):126-32. doi: 10.1097/NMD.0b013e3181961d8e. PMID 19214048
- [Background] Yesavage JA, Kinoshita LM, Kimball T, Zeitzer J, Friedman L, Noda A, David R, Hernandez B, Lee T, Cheng J, O'hara R. Sleep-disordered breathing in Vietnam veterans with posttraumatic stress disorder. Am J Geriatr Psychiatry. 2012 Mar;20(3):199-204. doi: 10.1097/JGP.0b013e3181e446ea. PMID 20808112
- [Background] Krakow B, Melendrez D, Johnston L, Warner TD, Clark JO, Pacheco M, Pedersen B, Koss M, Hollifield M, Schrader R. Sleep-disordered breathing, psychiatric distress, and quality of life impairment in sexual assault survivors. J Nerv Ment Dis. 2002 Jul;190(7):442-52. doi: 10.1097/00005053-200207000-00004. PMID 12142845
- [Background] Krakow B, Lowry C, Germain A, Gaddy L, Hollifield M, Koss M, Tandberg D, Johnston L, Melendrez D. A retrospective study on improvements in nightmares and post-traumatic stress disorder following treatment for co-morbid sleep-disordered breathing. J Psychosom Res. 2000 Nov;49(5):291-8. doi: 10.1016/s0022-3999(00)00147-1. PMID 11164053
- [Background] Webber MP, Lee R, Soo J, Gustave J, Hall CB, Kelly K, Prezant D. Prevalence and incidence of high risk for obstructive sleep apnea in World Trade Center-exposed rescue/recovery workers. Sleep Breath. 2011 Sep;15(3):283-94. doi: 10.1007/s11325-010-0379-7. Epub 2010 Jul 1. PMID 20593281
- [Background] van Liempt S, Westenberg HG, Arends J, Vermetten E. Obstructive sleep apnea in combat-related posttraumatic stress disorder: a controlled polysomnography study. Eur J Psychotraumatol. 2011;2. doi: 10.3402/ejpt.v2i0.8451. Epub 2011 Dec 26. PMID 22893807
- [Background] Kinoshita LM, Yesavage JA, Noda A, Jo B, Hernandez B, Taylor J, Zeitzer JM, Friedman L, Fairchild JK, Cheng J, Kuschner W, O'Hara R, Holty JE, Scanlon BK. Modeling the effects of obstructive sleep apnea and hypertension in Vietnam veterans with PTSD. Sleep Breath. 2012 Dec;16(4):1201-9. doi: 10.1007/s11325-011-0632-8. Epub 2011 Dec 23. PMID 22193972
- [Background] Ahmadi N, Hajsadeghi F, Mirshkarlo HB, Budoff M, Yehuda R, Ebrahimi R. Post-traumatic stress disorder, coronary atherosclerosis, and mortality. Am J Cardiol. 2011 Jul 1;108(1):29-33. doi: 10.1016/j.amjcard.2011.02.340. Epub 2011 Apr 29. PMID 21530936
- [Background] Sharafkhaneh A, Giray N, Richardson P, Young T, Hirshkowitz M. Association of psychiatric disorders and sleep apnea in a large cohort. Sleep. 2005 Nov;28(11):1405-11. doi: 10.1093/sleep/28.11.1405. PMID 16335330
- [Background] Bixler EO, Vgontzas AN, Ten Have T, Tyson K, Kales A. Effects of age on sleep apnea in men: I. Prevalence and severity. Am J Respir Crit Care Med. 1998 Jan;157(1):144-8. doi: 10.1164/ajrccm.157.1.9706079. PMID 9445292
- [Background] El-Solh AA, Ayyar L, Akinnusi M, Relia S, Akinnusi O. Positive airway pressure adherence in veterans with posttraumatic stress disorder. Sleep. 2010 Nov;33(11):1495-500. doi: 10.1093/sleep/33.11.1495. PMID 21102991
- [Background] Weathers F, Litz B, Herman D, et al. (October 1993). The PTSD Checklist (PCL): Reliability, validity, and diagnostic utility. Paper presented at the Annual Convention of the International Society for Traumatic Stress Studies, San Antonio, TX.
- [Background] Yeager DE, Magruder KM, Knapp RG, Nicholas JS, Frueh BC. Performance characteristics of the posttraumatic stress disorder checklist and SPAN in Veterans Affairs primary care settings. Gen Hosp Psychiatry. 2007 Jul-Aug;29(4):294-301. doi: 10.1016/j.genhosppsych.2007.03.004. PMID 17591505
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Derived] Orr JE, Smales C, Alexander TH, Stepnowsky C, Pillar G, Malhotra A, Sarmiento KF. Treatment of OSA with CPAP Is Associated with Improvement in PTSD Symptoms among Veterans. J Clin Sleep Med. 2017 Jan 15;13(1):57-63. doi: 10.5664/jcsm.6388. PMID 27707436